CLINICAL TRIAL: NCT03084432
Title: Assessment of Bone Mineral Content for Preterm Neonates Treated With Caffeine Using Dual Energy X-ray Absorptiometry : an Observational Study
Brief Title: Effect of Caffeine on Preterm Infants' Bone Mineral Content
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Ismail, Assistant Professor, Ain Shams University
Other Study IDs: 16246
Record Dates: First submitted 2017-03-10; First posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Osteopenia (Disorder); Apnea of Prematurity
Keywords: caffeine; bone mineral content
MeSH Terms: conditions — Bone Diseases, Metabolic; Apnea | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- caffeine group: 22 preterm infants received caffeine (starting from day 2 of life and received for more than 7 days) for apnea prophylaxis or treatment according to protocol of Ain Shams University neonatal intensive care unit [apnea prophylaxis for preterm ≤32 weeks gestation and apnea treatment for those 33 or 34 weeks gestation]. Dual Energy X-ray Absorptiometry was done 5th-6th week post-natal age
  Interventions: Diagnostic Test: Dual Energy X-ray Absorptiometry
- control group: 20 preterm infants for whom caffeine was not given, either it was not indicated, not available or parents refused its use.Dual Energy X-ray Absorptiometry was done 5th-6th week post-natal age
  Interventions: Diagnostic Test: Dual Energy X-ray Absorptiometry

INTERVENTIONS:
Diagnostic Test: Dual Energy X-ray Absorptiometry — Dual Energy X-ray Absorptiometry done for both studied groups

SUMMARY:
The primary objective was to determine whether caffeine therapy is associated with decreases bone mineral content using dual energy x-ray absorptiometry. Secondary objectives were to determine whether caffeine therapy is associated with increased incidence of nephrocalcinosis or bone fracture.

ELIGIBILITY:
Inclusion Criteria:

Preterm infants with gestational age of 34 weeks or less consecutively admitted to the neonatal intensive care unit

Exclusion Criteria:

Renal or endocrinal diseases Congenital anomalies Suspected chromosomal aberrations Receiving diuretics or steroid therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: preterm neonates
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
effect of caffeine therapy on bone mineral content using Dual Energy X-ray Absorptiometry | 5-6 weeks
  Whole Body Scanner, Pencil beam, regions: antro-posterior Spine, Lateral, Hip, Forearm/ Hand, Ortho Femur Speed: Up To 76mm Per Sec., Scan Times (min): antro-posterior Spine-2, Lateral-12, Hip-4, Forearm-1, Femur-4 Pentium II Computer System, Windows O/S, Lunar Software 15" Hi-Resolution Monitor, Auto Centering Laser Guide, Data Analysis: Auto Analysis Software, Smart Scan, Auto Position. Weight and length were measured and recorded. During the scan an infant was placed on the scanning table with the head at the marked start line, assuring that the position was the same for all subjects. The study was carried out with the infants sleeping without sedation. The infants were placed supine and were restrained with a cotton blanket. To induce sleep, infants were fed a few minutes prior to the study. When image quality was poor due to movement of the infant or to other causes the measurement at that time point was not included for analysis.

IPD SHARING:
Plan to Share IPD: No